CLINICAL TRIAL: NCT06530680
Title: Upper Extremity Function, Activity, Participation, and Engagement Before and After Hippotherapy in Children With Autism Spectrum Disorder and/or Cerebral Palsy
Brief Title: Upper Extremity Function Before and After Hippotherapy in Children With Autism Spectrum Disorder and/or Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: Nationwide Children's Hospital (Other); University of Montana (Other)
Responsible Party: Principal Investigator, Jill Heathcock, Professor, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020B0434
Record Dates: First submitted 2024-07-24; First posted 2024-07-31 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Autism Spectrum Disorder; Cerebral Palsy
MeSH Terms: conditions — Autism Spectrum Disorder; Cerebral Palsy | interventions — Equine-Assisted Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physical therapy incorporating hippotherapy and the equine environment (Experimental): Four 1 hour Hippotherapy treatments per week for four weeks.
  Interventions: Behavioral: Hippotherapy
- Waitlist Control (No Intervention): A waitlist control that will receive hippotherapy intervention (four 1 hour Hippotherapy treatments per week for four weeks.) Four weeks later than the 'Physical therapy incorporating hippotherapy and the equine environment' Group.

INTERVENTIONS:
Behavioral: Hippotherapy — Two 1-hour sessions of hippotherapy for eight weeks.
  Arms: Physical therapy incorporating hippotherapy and the equine environment

SUMMARY:
The goal of this feasibility trial is to learn if hippotherapy and physical therapy in the equine environment can be used to improve upper extremity function in children with cerebral palsy or autism spectrum disorder who present with motor delay or impairment in the upper extremities. The main questions it aims to answer are:

Can the upper extremity-focused treatment using hippotherapy and the equine environment be delivered to fidelity?

Is the treatment acceptable to participants and therapists?

Is the randomized-controlled trial protocol feasible to scale to a larger study, including recruitment and retention rates and suitability of selected outcome measures?

If there is a comparison group: Researchers will compare participants receiving treatment to a waitlist control to see if participants are retained in the control group and if differences are detected between the control and treatment groups on selected outcome measures.

DETAILED DESCRIPTION:
Intervention. Participants will receive 4 weeks of hippotherapy, 4 × 1-hour sessions per week, for a total of 16 hours of intervention. If the participants miss a session, make-up sessions will be offered, scheduled, and tracked.51

Hippotherapy: The hippotherapy intervention will be delivered at Dreams on Horseback in central Ohio using Professional Association of Therapeutic Horsemanship (PATH) Intl. standards. Participants will be mounted on a horse for at least 30 minutes of the 1-hour session. Activities for the remaining time include grooming and tacking of the horses, mounting, and dismounting. A herd of 9 horses will be used for hippotherapy sessions. There will be 2 volunteers assisting with every session: one to lead the horse, and one to walk alongside the participant opposite the treating therapist. Dreams on Horseback has a part-time Volunteer Coordinator who currently schedules 154 volunteers for 22 hours of equine-assisted activities per week (Monday - Saturday). Activities will include various positions on the horse such as sitting and quadruped (weight bearing through the upper extremities and knees), as well as reaching and throwing, controlling the horse with the reins, and riding the horse at a walk and a trot as is suggested by PATH Intl. Standards. Using the observation protocol in the preliminary data section, one researcher will video record one hippotherapy session each week and document the therapeutic activities performed. A second researcher will score 20% of the sessions to assure reliability of >90%. Categories expected based on preliminary data are transitions, ground poles, directional changes, reaches outside of base of support, reaches, weight bearing through upper extremities, using reins, holding upper extremities off of the horse, position on the horse (with or without stirrups, standing, sitting, posting), and kicking/squeezing the horse with legs. This analysis will allow the investigators to quantify the dose of hippotherapy, focus on the impact of therapeutic targets to the upper extremities, and allow the investigators to evaluate adherence to the hippotherapy protocol.

Treating Therapists: All treating therapists will be licensed PTs and will have completed at least the AHA Level I Hippotherapy Treatment Principles.

Since the goal of pilot studies is not to test efficacy, no inferential statistics are proposed. The investigators will analyze questions pertaining to 1) the recruitment success of children with CP+ASD ages 5-15; 2) whether participants adhere to what they are asked to do during the pilot RCT; and 3) if the treatment can be successfully delivered per protocol. The investigators will describe the number of potential participants screened per month; the number enrolled per month; the average time delay from screening to enrollment; and the average time to enroll enough participants for 2 groups. Treatment-specific retention and attrition rates for hippotherapy, including the reasons for dropouts, and treatment-specific fidelity rates, including a measure of dose of hippotherapy and upper extremity activities, will be described.

ELIGIBILITY:
Inclusion Criteria:

* Children age 6 to 17
* Diagnosis of Cerebral Palsy with Gross Motor Functional Classification System (GMFCS) Level I, II, or III with upper extremity affected Cerebral Palsy and/or Autism Spectrum Disorder
* Able to follow simple verbal instructions in English
* Able to tolerate sitting on a horse continuously for 30 minutes

Exclusion Criteria:

* Fear of or aversion to horses
* Weight over 200 lb
* Lacking independent head control (GMFCS level IV and V)
* Both parents unable to speak and read English

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2021-06-14 (Actual); Primary Completion 2023-02-03 (Actual); Study Completion 2023-02-03 (Actual)

PRIMARY OUTCOMES:
Reach-and grasp protocol | 1 week pre- and post- 4-week waitlist control period and within 1 week pre- and post- 4-week treatment period.
  Reach-and-grasp protocol: Participants were recorded while performing a reach-to-drink task. For each trial, participants were instructed: "Reach for the bottle, pick it up, pretend to take a drink, return the bottle to the marked position on the table, and return your hand to the start position. Do this twice." Movement of the upper extremities was recorded from reflective markers on the hands, wrists, elbows, shoulders, and sternum by a 10-camera VICON Motion Capture system at 120 Hz and filtered at 4 Hz with a low-pass Butterworth filter.
PEM-CY | 1 week pre- and post- 4-week waitlist control period and within 1 week pre- and post- 4-week treatment period
  Participation and Environment Measure for Children and Youth; higher scores mean better; participation scores range 0-7, involvement scores range 1-5.
PRIME-O | 1 time per week during the 4-week intervention period
  Pediatric Rehabilitation Intervention Measure of Engagement - Observation; higher scores = more engaged; score range = 0-40 (0-4 per item)
PRIME-SP | 1 time per week during the 4-week intervention period
  Pediatric Rehabilitation Intervention Measure of Engagement - Service Provider; not scaled
Enjoy | 1 time per week during the 4-week intervention period
  Self-report measure of enjoyment of an activity. The scale has 25 statements that respondents rate on a 7-point Likert scale the degree to which they agree or disagree with each statement. There are 5 sections of the measure that cover different components of enjoyment: pleasure, relatedness, competence, challenge/improvement, and engagement. higher scores = more enjoyment; scores range 1-7 per item.
VABS | 1 week pre- and post- 4-week waitlist control period and within 1 week pre- and post- 4-week treatment period
  Vineland Adaptive Behavior Scale 2nd Edition; high scores mean better; Adaptive Behavior Composite standard score range: 20-160.
CAPE/PAC | 1 week pre- and post- 4-week waitlist control period and within 1 week pre- and post- 4-week treatment period
  Child Assessment of Participation and Enjoyment / Preference for Activities in Children; higher scores mean better; score range CAPE = 55-275 (1-5 per item), PAC = 55-165 (1-3 per item)

CONTACTS AND LOCATIONS:
Locations (1):
- The Ohio State University, Columbus, Ohio, United States